CLINICAL TRIAL: NCT00339742
Title: Gastric and Esophageal Malignancies in Northern Iran (GEMINI): Phase I: Case-Control Study
Brief Title: Stomach and Esophageal Cancers in Northern Iran
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903146; 03-C-N146; NCT00544843 (obsolete NCT alias); NCT01338207 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Esophageal Cancer
Keywords: Esophageal Cancer; Case-Control Study; Environmental Risk Factors; Genetic Risk Factors
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood, hair, nails

GROUPS / COHORTS (3):
- Clinic Referral controls: Controls referred by the endoscopy clinic
- Esophageal Cancer cases: Histologically confirmed squamous cell cancer of the esophagus
- Neighborhood controls: Controls recruited from the neighborhood

SUMMARY:
This study, sponsored jointly by the National Cancer Institute and the Tehran University of Medical Sciences, will explore the causes of cancers of the stomach and esophagus (the tube that runs between the mouth and the stomach) in Northern Iran. This is a unique area of study for the following reasons:

* Some of the highest rates of esophageal cancer in the world have been reported in northeastern Iran 109 cases per 100,000 men and 175 cases per 100,000 women each year about 40 times higher than the rates of this cancer in the United States.
* In this area of Iran, unlike most areas of the world, the disease affects more women than men.
* Within 300 miles along the southern border of the Caspian Sea, the rates fall to 10 cases per 100,000 people per year.

The high rates of disease in this area, the unique geographic distribution of cases, and the exceptionally high rate in women make Northern Iran a promising site for studying esophageal and stomach cancers.

Patients 30 years of age and older who are referred to the upper gastrointestinal disease Atrak Clinic in Gonbad, Golestan Province, Iran, with suspected esophageal cancer may be eligible for this study. In addition, control subjects 30 years of age and older with certain specified diseases will be recruited from patients referred to four hospitals in Gonbad and to the Taleghani Clinic. After giving informed consent, all participants will undergo the following procedures:

* Interviews, including questions about age, ethnicity, education, and other demographic data; habits, such as tobacco, opium, and alcohol consumption; personal and family medical history; diet, with special attention to food preservation, cooking methods, and drinking water; physical activity; occupational and residential history; body measurements; signs and symptoms of upper gastrointestinal disease; oral hygiene; animal contact; transfusion history; and family socioeconomic status.
* Blood draw (15 milliliters, or 1 tablespoon) for genetic and chemical testing for markers that may predict who gets the disease.
* Hair and nail sampling to identify minerals or compounds whose exposure may be related to esophageal cancer.
* Endoscopy to evaluate the health of the esophagus and stomach. This test will be performed on all case patients and on control participants who give their permission. Before the examination, the subject will swallow a liquid that numbs the throat and may be given a medicine through a vein to promote drowsiness. The subject will then swallow a tube (endoscope) through which the doctor can look at the esophagus and stomach and take samples of tissue to look for disease. The tissue samples will be examined microscopically and will then be stored for possible future genetic or other testing related to diagnosing or determining the risk of esophageal cancer.

DETAILED DESCRIPTION:
This case-control study (the first phase of the GEMINI project) is primarily focused on exploring the etiology (etiologies) of squamous cell carcinoma of the esophagus in northern Iran.

Esophageal and gastric cancers, together, are responsible for more than 1,000,000 annual deaths in the world. In 1996, cancers of the stomach and esophagus ranked first and second respectively, among the most frequent cancers in Iran, excluding skin cancers. Some of the highest incidence rates for esophageal cancer in the world have been reported in Northeastern Iran, in Northern Gonbad, with Age Standardized Rates (ASR) of 109/100,000 in men and 175/100,000 in women (1). These rates are approximately 40 times higher than those seen in the US. In this area, unlike most areas of the world, the incidence is higher in women than in men. Additionally, within 300 miles along the southern border of Caspian Sea, the rates fall to 10/100,000. The highest rates of EC in the world, a unique geographical distribution of cases, and an exceptionally high rate among women all make Northern Iran a very intriguing site for studying this disease.

An upper-GI referral clinic (Atrak Clinic) has already been established in Gonbad, Golestan Province, and DDRC researchers have conducted feasibility studies in this clinic. For the case-control study, local internists and other health system workers will refer suspected cases of esophageal cancer to the Clinic. All such patients will undergo endoscopy and biopsy for ascertainment of diagnosis. Patients who have histologically confirmed esophageal squamous cell carcinoma of the esophagus and consent to join the study will be enrolled as cases. There will be two control groups in this study, one selected from the neighborhood of case subjects and one from the patients referred to Atrak Clinic who do not have cancer. The neighborhood control group will serve as the primary control group. Both the cases and the controls will be interviewed and undergo collection of biological specimens including blood, hair and nails. Free (and optional) endoscopy will also be offered to the neighborhood controls. A four-year accrual of 300 cases, 600 neighborhood controls and 300 clinic controls is expected.

Environmental risk factors (including life-style, habits, and nutritional status) will be assessed through questionnaires and objective measurements in biological specimens. The role of genetic polymorphisms will be studies using genomic DNA from cases and controls. A subset of samples collected from cases and controls will be used to evaluate gene expression patterns, using microarray analysis, differences in serum protein patterns, using SELDI analysis.

ELIGIBILITY:
* INCLUSION CRITERIA:

Cases:

Cases will be recruited and studied in Atrak Clinic, in Gonbad City.

All patients referred to Atrak Clinic suspected to have EC.

Patients 30 years of age or above from Gonbad, Minodasht, Kalaleh, Ramyan, Azad-Shahr, Maraveh-Tappeh, and the surrounding villages who have a histopathological diagnosis confirming ESCC and who consent to join the study will be enrolled as cases.

Controls:

Controls will be recruited into one of the four hospitals of the city (Shohada, Motahary, Khatam, and Borzouieh), and in major referral outpatient clinic (Taleghani Clinic).

Controls will be selected from the patient 30 years of age or above who are referred to the four hospitals of the city and Taleghani Clinic.

Only patients referred for certain diseases will be selected as controls.

EXCLUSION CRITERIA:

Controls:

No association with tobacco or alcohol consumption, which are the main known risk factors for esophageal cancer (such as lung cancer, cardiovascular disease.

Not causing major changes in diet or life-style for a long time (such as major GI diseases, chronic malignancies, diabetes).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have histologically confirmed esophageal squamous cell carcinoma of the esophagus and consent to join the study were enrolled as cases. There were two control groups in this study, one selected from the neighborhood of case subjects and one from the patients referred to Atrak Clinic who do not have cancer. The neighborhood control group served as the primary control group.
Sampling Method: Non-Probability Sample
Enrollment: 1163 (Actual)
Dates: Start 2003-03-25 (Actual); Primary Completion 2010-03-26 (Actual); Study Completion 2020-02-13 (Actual)

PRIMARY OUTCOMES:
Esophageal Cancer | At diagnosis
  Patients who have histologically confirmed esophageal squamous cellcarcinoma of the esophagus and consent to join the study will be enrolled as cases.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Abnet, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Digestive Disease Research Center, Tehran University of Medical Sciences, Tehran, Iran

REFERENCES:
- [Background] Abnet CC, Kamangar F, Islami F, Nasrollahzadeh D, Brennan P, Aghcheli K, Merat S, Pourshams A, Marjani HA, Ebadati A, Sotoudeh M, Boffetta P, Malekzadeh R, Dawsey SM. Tooth loss and lack of regular oral hygiene are associated with higher risk of esophageal squamous cell carcinoma. Cancer Epidemiol Biomarkers Prev. 2008 Nov;17(11):3062-8. doi: 10.1158/1055-9965.EPI-08-0558. PMID 18990747
- [Background] Islami F, Pourshams A, Nasrollahzadeh D, Kamangar F, Fahimi S, Shakeri R, Abedi-Ardekani B, Merat S, Vahedi H, Semnani S, Abnet CC, Brennan P, Moller H, Saidi F, Dawsey SM, Malekzadeh R, Boffetta P. Tea drinking habits and oesophageal cancer in a high risk area in northern Iran: population based case-control study. BMJ. 2009 Mar 26;338:b929. doi: 10.1136/bmj.b929. PMID 19325180
- [Background] Islami F, Kamangar F, Nasrollahzadeh D, Aghcheli K, Sotoudeh M, Abedi-Ardekani B, Merat S, Nasseri-Moghaddam S, Semnani S, Sepehr A, Wakefield J, Moller H, Abnet CC, Dawsey SM, Boffetta P, Malekzadeh R. Socio-economic status and oesophageal cancer: results from a population-based case-control study in a high-risk area. Int J Epidemiol. 2009 Aug;38(4):978-88. doi: 10.1093/ije/dyp195. Epub 2009 May 4. PMID 19416955